CLINICAL TRIAL: NCT01659112
Title: Does Core Stabilization Enhance Neuromuscular Control and Functional Status of the Upper Extremity?
Brief Title: Effects of Core Stabilization Approach on Patients With Upper Extremity Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cigdem Ayhan, Lecturer, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 010T03102001
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-08

CONDITIONS: Upper Extremity Injuries
Keywords: core stabilization, upper extremity, kinetic chain, movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stabilization Group (Experimental): A core stabilization plus traditional upper extremity rehabilitation approach was performed.
  Interventions: Other: Core Stabilization; Other: Traditional upper extremity rehabilitation
- Control Group (Active Comparator): A traditional upper extremity rehabilitation-only approach was performed.
  Interventions: Other: Traditional upper extremity rehabilitation

INTERVENTIONS:
Other: Core Stabilization — A 6-week (3 days a week) exercise intervention including progressive core exercises was performed.
  Arms: Stabilization Group
Other: Traditional upper extremity rehabilitation — A 6-week (3 days a week) exercise intervention of the injured joint based on the recovery process was performed.

SUMMARY:
The purpose of the study is to determine the effects of the addition of core stabilization exercises to a traditional upper extremity rehabilitation program in upper extremity injuries.

DETAILED DESCRIPTION:
Abnormal movement patterns are one of the most challenging problems during rehabilitation of the patients with upper extremity injuries. They usually decrease the functional status of the upper extremity and prevent isolated muscle activations. Dysfunction of the kinetic chain system plays an important role in the development of these movement patterns. Thus, multi-segmental rehabilitation strategies has recently gained considerable importance in upper extremity rehabilitation. Core stabilization is one of the most popular rehabilitation approaches preferred to enhance functional stability of the kinetic chain system and dynamic postural alignment during activities. The purpose of this study is to determine the effects of core stabilization approach on functional status of the upper extremity and the amount of abnormal movement patterns. In addition, the factors affecting the abnormal movement patterns will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic distal segment injuries (elbow and wrist)
* Patients in their subacute stage.

Exclusion Criteria:

* Multiple joint problems
* Bilateral extremity problems
* Reflex sympathetic dystrophy
* Trunk and lower extremity problems
* Non-union fractures
* Malignant ans systemic diseases

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Upper extremity functional status | 30 minutes
  Pain Range of motion Endurance Fatigue severity DASH

SECONDARY OUTCOMES:
Measurement of abnormal movement patterns | 1 hour
  Video analysis during two daily living activities (hand to mouth and opening doorknob) was recorded for both injured and uninjured extremity before and after the intervention.

OTHER OUTCOMES:
Trunk muscle strength | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Ünal, PhD, Prof, Study Director — Hacettepe University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation
Locations (1):
- Hacettepe University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Ayhan C, Unal E, Yakut Y. Core stabilisation reduces compensatory movement patterns in patients with injury to the arm: a randomized controlled trial. Clin Rehabil. 2014 Jan;28(1):36-47. doi: 10.1177/0269215513492443. Epub 2013 Jul 3. PMID 23823711